CLINICAL TRIAL: NCT07142551
Title: Supraphysiologic Testosterone Priming Induces Darolutamide Extended Response Via Modulation of ANdrogen Receptor (the SPIDERMAN Trial)
Brief Title: Supraphysiologic Testosterone Priming Induces Darolutamide Extended Response
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J2564; IRB00509292 (Other: JHM IRB)
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone 17 beta-cypionate; Gonadotropin-Releasing Hormone; Triptorelin Pamoate; luprolide acetate gel depot; Leuprolide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; relugolix; darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lead-In Phase - ADT with an LHRH agonist or antagonist (Experimental): Eligible patients will initiate combined androgen deprivation therapy (ADT) with an LHRH agonist or antagonist (e.g. Eligard, Zoladex, Lupron, Orgovyx) in combination with standard dose darolutamide (600 mg twice daily) for a total of 6 months. After this initial "lead-in" phase, patients who have clinical or radiographic progression or do not have at least a ≥50% decline in PSA will remain on combined androgen deprivation and discontinue study.
  Interventions: Drug: Luteinizing hormone-releasing hormone (LHRH) analogue; Drug: Darolutamide
- Bipolar Androgen-based Therapy (BAT) Cycle (Experimental): Patients with ≥50% decline in PSA will discontinue combined androgen deprivation and will receive intermittent intramuscular testosterone cypionate (T) at a dose of 400 mg every 4 weeks for a total of 3 injections while on a BAT cycle (12 weeks).
  Interventions: Drug: Testosterone cypionate
- Darolutamide Cycle (Experimental): Patient will proceed to a cycle off BAT and start darolutamide alone at 600 mg twice daily for 12 weeks. Patients will continue with alternating cycles of BAT or darolutamide (without ADT) until clinical or radiographic progression.
  Interventions: Drug: Darolutamide

INTERVENTIONS:
Drug: Testosterone cypionate — Intermittent intramuscular testosterone cypionate (T) at a dose of 400 mg every 4 weeks.
  Other Names: Depo-Testosterone
  Arms: Bipolar Androgen-based Therapy (BAT) Cycle
Drug: Luteinizing hormone-releasing hormone (LHRH) analogue — Eligible patients will initiate combined androgen deprivation therapy (ADT) with an LHRH agonist or antagonist (e.g. Eligard, Zoladex, Lupron, Orgovyx) in combination with standard dose darolutamide (600 mg twice daily) for a total of 6 months.
  Other Names: Trelstar; Eligard; Lupron; Degarelix; Relugolix
  Arms: Lead-In Phase - ADT with an LHRH agonist or antagonist
Drug: Darolutamide — 600 mg twice daily during the lead-in phase and on darolutamide cycle.
  Other Names: Nubeqa
  Arms: Darolutamide Cycle; Lead-In Phase - ADT with an LHRH agonist or antagonist

SUMMARY:
The objective of this study is to determine the safety and clinical effects of alternating pharmacologic (i.e. supraphysiologic) testosterone therapy with darolutamide in men with metastatic prostate cancer as first line hormonal therapy. Correlative studies will be conducted to assess the effect of alternating therapy on quality of life, gene expression and metabolic changes associated with alternating therapy.

DETAILED DESCRIPTION:
This research is being done to determine if alternating high dose testosterone and prevent the development of resistance to hormone therapy. It is also being done to determine if this alternating therapy can decease the side effects of hormone therapy and improve the participant's quality of life.

Right now, patients who develop metastatic prostate cancer are treated with medications that block testosterone effects as first-line therapy. Eventually, the testosterone blocking therapies become ineffective and the tumor begins to grow. The investigaors call this phase of the disease castrater-resistant prostate cancer (CRPC). Previous research has shown that prostate cancer cells can eventually adapt to low testosterone conditions produced by hormone therapy and begin to grow again. The investigators have learned that these resistant prostate cancer cells can killed by high levels of testosterone followed by a rapid drop to low testosterone levels. The investigators call this treatment bipolar androgen therapy (BAT) because the investigators are going from the polar extremes of high and low testosterone in the blood every 28 days. The investigators have tested this idea in previous studies by giving injections of high doses of testosterone to patients with CRPC. In these trials, the investigators saw that BAT was safe. BAT produced decreases in PSA levels and decreases in tumor size in some patients. After treatment with BAT, many patients had an improved response to the testosterone-blocking drug enzalutamide. The drug used in this study, darolutamide, is similar to enzalutamide. Both drugs are considered to be antiandrogens that block effects of testosterone within the prostate cancer cells.

The investigators also did a study called the BATMAN study in patients with mHSPC. These patients received alternating therapy with high dose testosterone and ADT as first line therapy. In this study, alternating testosterone and ADT was found to be safe. In this study, more patients remained sensitive to hormone therapy after 18 months than the investigators would have expected with ADT alone.

In this study, the investigators would like to see if improvement on these results and decrease hormonal side effects when the investigators give testosterone in sequence with darolutamide.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Performance status ≤2.
* Documented histologically confirmed adenocarcinoma of the prostate.
* Baseline PSA ≥1.0 ng/ml.
* No prior androgen deprivation therapy (i.e. surgical castration LHRH agonist, LHRH antagonist) as treatment for biochemically recurrent or metastatic disease (may have received neoadjuvant, concurrent and/or adjuvant AD therapy in the context of definitive radiation therapy if it was administered ≥ 1 year prior to recurrence).
* No prior treatment with ARPI (abiraterone, enzalutamide, darolutamide) for biochemically recurrent or metastatic prostate cancer. Neoadjuvant, concurrent and/or adjuvant ARPI +/- ADT is permitted if given in the context of definitive radiation therapy if it was administered ≥ 1 year prior to development of metastatic disease.
* Prior focal radiation treatment (e.g. SABR, Cyberknife) for oligometastatic disease is permitted if > 6 months. Patients must have evidence of metastatic disease in non-irradiated sites to be eligible for study.
* Evidence of rising PSA on two successive dates > 2 weeks apart.
* Evidence of metastatic disease on CT scan or bone scan performed with six weeks of screening.
* Patients with bone pain due to prostate cancer are eligible for trial but must be pain free at the end of the 6-month lead-in phase to be eligible to receive subsequent BAT.
* Patients with soft tissue lesions amenable to biopsy must agree to baseline and 6 months tumor biopsies to enroll in study.
* Acceptable liver function:

  1. Bilirubin < 2.5 times institutional upper limit of normal (ULN)
  2. AST (SGOT) and ALT (SGPT) < 2.5 times ULN
* Acceptable renal function:

  a. Serum creatinine < 2.5 times ULN
* Acceptable hematologic status:

  1. Absolute neutrophil count (ANC) > 1000 cells/mm3 (1.0 ×109/L)
  2. Platelet count > 100,000 platelet/mm3 (100 ×109/L)
  3. Hemoglobin > 9 g/dL.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* No prior treatment with chemotherapeutic regimens allowed.
* No prior treatment with Pluvicto or other PSMA-targeted agents is allowed.
* No prior treatment with Androgen Receptor targeted investigational agents is permitted.
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
* Evidence of disease that, in the opinion of the investigator, would put the patient at risk from testosterone therapy (e.g. femoral metastases with concern over fracture risk, spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction).
* Requires urinary self-catheterization for voiding due to obstruction secondary to prostatic enlargement well-documented to be due to prostate cancer or benign prostatic hyperplasia (BPH). Patients with indwelling Foley or suprapubic catheter for obstructive symptoms are eligible.
* Active uncontrolled infection.
* Any condition or mental impairment that may compromise the ability to give informed consent, patient's safety or compliance with study requirements as determined by the investigator.
* Patients receiving anticoagulation therapy with Warfarin or Coumadin are not eligible for study. Patients on non-coumadin anticoagulants (Lovenox, Eliqis, Xarelto, etc.) are eligible for study. Patients on Coumadin who can be transitioned to non-coumadin anticoagulants prior to starting study treatments will be eligible.
* Hematocrit >51%, untreated severe obstructive sleep apnea, uncontrolled or poorly controlled heart failure [per Endocrine Society Clinical Practice Guidelines (34)]
* Patients allergic to sesame seed oil or cottonseed oil are excluded.
* Major surgery as determined by the treating physician within 3 weeks before screening, or has not fully recovered from prior surgery (i.e., unhealed wound). Note: subjects with planned procedures (minor surgery with local anesthesia), colonoscopy under anesthesia may participate.
* Abnormal cardiac function as manifested by NYHA (New York Heart Association) class III or IV heart failure or history of a prior myocardial infarction (MI) within the last five years prior to enrollment in the study.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects free of Clinical or radiographic free progression | 24 months from Day 1 (start of treatment)
  Percent of subjects are free of clinical or radiographic progression at 24 months from initiation of treatment

SECONDARY OUTCOMES:
Percent of patients who achieve Complete PSA response at end of in lead-in phase | 6 months from Day 1 (start of treatment)
  Percent of patients who achieve a complete PSA response (i.e. serum PSA <0.2 ng/ml) at end of in lead-in phase.
Percent of patients who achieve Complete PSA response with darolutamide treatment | 36 months from Day 1 (start of treatment)
  Percent of patients who achieve a complete PSA response (i.e. serum PSA <0.2 ng/ml) over the course of treatment with darolutamide.
Number of patients with Clinical or Radiographic progression free survival | 6 years from Day 1 (start of treatment)
  Number of patients with clinical or radiographic progression free survival while on the study.
Overall Survival | 6 years from Day 1 (start of treatment)
  Number of months from the start of study treatment in the lead-in phase to death due to any cause, will be summarized using Kaplan-Meier method
Objective Response to darolutamide | 1 year from Day 1 (start of treatment)
  Number of patients who have complete response or partial response according to RECIST 1.1 criteria, among those with measurable disease at baseline, with darolutamide treatment following BAT.
Response in patients with high volume (CHAARTED criteria) vs. low volume disease | 3 years from Day 1 (start of treatment)
  Number of patients who have complete response or partial response according to RECIST 1.1 criteria, among those with measurable disease at baseline, with high volume disease vs those with low volume disease.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events | 3 years from Day 1 (start of treatment)
  Measured by the number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Quality of Life as assessed by the Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale | 2.5 years from Day 1 (start of treatment)
  Quality of life over time based on the FACIT-Fatigue. The Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function. The total score ranges between 0 and 52, with higher scores denoting less fatigue.
Quality of Life as assessed by the Short Form-36 (SF-36) | 2.5 years from Day 1 (start of treatment)
  Quality of life over time based on the SF-36 survey. Short Form 36 (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. Score range 0-100, lower scores represent more physical function disability, while higher scores represent less disability.
Quality of Life as assessed by the International Index of Erectile Function (IIEF) | 2.5 years from Day 1 (start of treatment)
  Quality of life over time based on the IIEF survey. The 15-question IIEF Questionnaire is a validated, multidimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. A scale of 0-5, is awarded to each of the 15 questions with a total score range 0-75 that examines the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. Higher scores represent more severe erectile dysfunction, while lower scores represent less erectile dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No